CLINICAL TRIAL: NCT06590818
Title: The Effect of Body Mass Index on Short-term Results of HTO for Treatment of OA With Varus Knee in Upper Egypt Population
Brief Title: The Effect of Body Mass Index on Short-term Results of HTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahmed Ramadan Hammad
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Osteo Arthritis Knee; Varus Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- varus knee osteoarthritis Group (Experimental): About 50 patients had varus knee osteoarthritis underwent high tibial osteotomy (HTO)
  Interventions: Procedure: High tibial osteotomy (HTO

INTERVENTIONS:
Procedure: High tibial osteotomy (HTO — To investigate the effect of body mass index (BMI) on the early efficacy of high tibial osteotomy (HTO) in the treatment of varus knee osteoarthritis
  Other Names: Effect of body mass index (BMI)

SUMMARY:
The knee joint plays a major role in weight transmission of the body in day-to-day activities. The biomechanics of the knee and malalignment in lower limb anatomy are major risk factors for chronic knee pain, leaving Total Knee Arthroplasty (TKA) as the best and most successful option for patients with end-stage osteoarthritis (OA)

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative disease characterized by progressive joint damage.The knee is one of the joints most affected by this pathology, and it is estimated that 10% of men and 13% of women older than 60 years present it.It is characterized by pain, functional limitation, and reduction of quality of life.

Knee osteoarthritis (KOA) is a multi-etiological, chronic disabling disease that affects the entire knee joint, which is the most common site of involvement in OA. KOA is classified as primary or secondary depending on etiology. The pathogenesis of primary KOA is complex and involves numerous factors, such as mechanical stress, inflammation, metabolism, immunity and genetics, with age, genetics, body weight, sex and race being risk factors.

Diagnosis of knee osteoarthritis can be confirmed based on clinical and/or radiological features. The potential of a progressive disease can be prevented or decreased by earlier recognition and correction of associated factors.Obesity and alignment especially varus malalignment are recognized factors of a progressive disease. Both non pharmalogical as well as pharmacological modalities of treatment are useful in managing the symptoms of knee osteoarthritis. Surgery should be considered only in patients who do not respond to medical therapy.

Varus knee osteoarthritis is one of the most common knee diseases in clinical practice. Knee pain and limited range of motion seriously affect the patient's quality of life. However, there is need for further exploration into the prevention and treatment of postoperative complications following artificial joint replacement.

Osteotomy techniques such as high tibial osteotomy are primarily used for the treatment of KOA with varus and valgus deformities.

High body mass index is a risk factor for KOA. A previous study reported a 35% increase in KOA risk with every 5-unit increase in body mass index. This is primarily attributed to the fact that greater body weight increases the weight-bearing pressure of the knee joint, thereby increasing the probability of KOA

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for knee osteoarthritis and only have one knee
* No serious underlying medical disease
* Conservative treatment is ineffective and there is a willingness for surgery
* X-ray shows degeneration limited to the medial joint space (Ahlback grade ≥ grade II)
* Knee flexion range of motion > 90°, varus deformity < 15°, flexion contracture < 5°.
* Clinical examination shows intact anterior cruciate ligament and collateral ligament, tenderness point is limited to the medial joint space, and the lateral compartment and patellofemoral joint are intact.

Exclusion Criteria:

* knee osteoarthritis caused by infection, blood-related or autoimmune diseases.
* severe obesity (BMI>35 kg/m 2 ) or morbid obesity (obesity caused by diseases such as hypercortisolism and hypothyroidism, BMI≥30 kg/m 2 ).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Blood Loss (defined as blood loss ≥500 cc) | First 2 hours till 3 days after the operation
  Assessment of bleeding intraoperative and post operative by measuring Hemoglobin level and Hematocrit level pre and post operation.

SECONDARY OUTCOMES:
Knee Joint Function | Two hours after the operation
  Evaluated using HSS score, knee range of motion before and after the operation.
Assessment of Pain | Two hours after the operation
  Assessment of Pain by using VAS score for pain status

CONTACTS AND LOCATIONS:
Overall Officials: Maysara Abdelhaleem Bayuomy, Assist.Prof, Study Chair — Orthopedic &Trauma surgery Department, Faculty of medicine, Al-Azhar University, Assiut
Locations (1):
- Al-Azhar University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided